CLINICAL TRIAL: NCT02998944
Title: the Association Study of Constitution of Traditional Chinese Medicine and Common Diseases
Brief Title: The Study of CCTM and Common Diseases
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zihui Tang, Attending physician, Huashan Hospital
Other Study IDs: cctmcd
Record Dates: First submitted 2016-12-04; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension; Diabetes Mellitus; Chronic Obstructive Pulmonary Disease Moderate; Coronary Artery Disease; Obesity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Coronary Artery Disease; Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other:  — not any intervention for this study

SUMMARY:
This study aimed to explore the associations between constitutions of traditional Chinese medicine (TCM) and common disease (CD). A large-scale, community-based, cross-sectional study was performed to investigate the associations. A total of 3748 participants were available for analysis in this study. The assessment of constitution of TCM was based on recommendations of Association Chinese Medicine in China. In this study, the diagnosis of CD was based on self-reported medical history. The associations were analyzed using univariate and multivariable logistic regression (MLR).

DETAILED DESCRIPTION:
This study aimed to explore the associations between constitutions of traditional Chinese medicine (TCM) and common disease (CD). A large-scale, community-based, cross-sectional study was performed to investigate the associations. A total of 3748 participants were available for analysis in this study. The assessment of constitution of TCM was based on recommendations of Association Chinese Medicine in China. In this study, the diagnosis of CD was based on self-reported medical history. The associations were analyzed using univariate and multivariable logistic regression (MLR).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 30-90 years were recruited from rural and urban communities in Shanghai.

Exclusion Criteria:

* severity renal and liver function abnormal and pregnant woman

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A risk-factor study for constitution of TCM and chronic disease was conducted in a random sample of the Chinese population. Participants aged 30-90 years were recruited from rural and urban communities in Shanghai. More than 4,000 participants were invited to a screening visit between 2011 and 2013. Written consent was obtained from all patients before the study, which was performed in accordance with the ethical standards in the Declaration of Helsinki, and approved by the Medicine Ethical Committee of the Huashan Hospital. The exclusion criteria were 1) severity renal and liver function abnormal and 2) pregnant woman. A total of 3748 participants were available to data analysis.
Sampling Method: Probability Sample
Enrollment: 3748 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
hypertension | through study completion, an average of 2 year
  questionaire
diabetes mellitus | through study completion, an average of 2 year
  questionaire
coronary artery disease | through study completion, an average of 2 year
  questionaire
COPD | through study completion, an average of 2 year
  questionaire
Obesty | through study completion, an average of 2 year
  calculation from height and weight

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang P, Dong J, Zeng F, Tang Z. Analysis of the association between glucose profiles and beta-cell function for diabetic cardiovascular autonomic neuropathy in China. J Diabetes Investig. 2017 May;8(3):354-362. doi: 10.1111/jdi.12584. Epub 2016 Nov 25. PMID 27736036
- [Background] Lv Y, Zhou L, Tang Z, Dong J. Association and interaction analysis of diabetes mellitus and SCN10A for cardiovascular autonomic neuropathy in a Chinese population. Postgrad Med J. 2017 Jun;93(1100):344-348. doi: 10.1136/postgradmedj-2016-134202. Epub 2016 Oct 11. PMID 27729462